CLINICAL TRIAL: NCT03244449
Title: Identification and Validation of Myonectin, Myostatin and FGF-21 as Insulin Resistance Biomarkers in Colombian People
Brief Title: New IR Biomarkers (Myokines) in Colombian People
Status: Completed | Type: Observational
Sponsor: University of Los Andes, Columbia (Other)
Collaborators: The Administrative Department of Science, Technology and Innovation, Colciencias (Other); Universidad Militar Nueva Granada (Unknown)
Responsible Party: Principal Investigator, Carlos O Mendivil, Associate Professor, University of Los Andes, Columbia
Other Study IDs: 120465745008
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Insulin Resistance; Diabetes Mellitus, Type 2
Keywords: biomarker; insulin resistance; myokine; clamp
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No apply

SUMMARY:
Around the world, the prevalence of type 2 diabetes mellitus (T2DM) has been increasing since the last two decades, with approximately 347 million patients with diabetes by 2013 according to the World Health Organization (WHO). This pronounced increase is due to an increase in the prevalence of obesity, reduction in physical activity levels, accelerated urbanization and aging of the population. In Colombia, T2DM ranks fifth in the main morbidity and mortality causes, including only deaths caused directly and without adding the strong influence that T2DM has on cardiovascular disease mortality.

Insufficient tissue response to normal insulin concentrations, called insulin resistance, is one of the central pathophysiological mechanisms in the development of T2DM. However, there is currently no simple, practical, safe and reproducible method that allows the diagnosis or identification of insulin resistance, nor the follow-up to its evolution. At the moment, the gold standard for assessing the degree of insulin sensitivity or resistance is the "hyperinsulinemic-euglycemic clamp", a laborious technique, of high cost and high technical difficulty, requiring specialized personnel and hospitalization. Non-invasive methods based on mathematical regressions, such as the Homeostatic Model Assessment (HOMA-IR), are imperfect and widely variable, and have not been validated in the Latin American population, less Still Colombian.

Therefore, the development of new, easily obtainable quantitative tools for the diagnosis of insulin resistance is required. This requires not only the identification of new and better biomarkers, but also the determination of their diagnostic performance and operational characteristics.

This project will investigate 3 molecular targets (myokines), novel and easy to measure, with high probability of being good biomarkers of insulin resistance. The research will include validation of its association with insulin resistance measured by the reference method, as well as its measurement in apparently healthy individuals. Finally, operator-receiver characteristics of each test will be analyzed, in order to propose a cutoff point for the diagnosis of insulin resistance.

DETAILED DESCRIPTION:
The objectives of the project are: 1) To identify, within a group of 3 potential new biomarkers of insulin resistance, those that are significantly associated with the presence of this phenomenon in our population, 2) Establish, analyze and apply reference values for each one of these three biomarkers in Colombian population. 3) To evaluate the sensitivity, specificity, statistical C (operational performance), predictive values and likelihood ratios of each of the biomarkers studied for the diagnosis of insulin resistance versus a standard gold technique and 4) Different biomarkers evaluated, in order to select the best one (s) for clinical use, as well as to propose a cutoff point for detection of insulin resistance for each of them.

Methodology: A cross-sectional, diagnostic test evaluation study will be conducted, including apparently healthy Adults of both sexes, with ages between 35 and 65 years, coming from Bogotá, without any significant comorbidity.

As initial evaluation will be carried out measurement of height, weight, percentage of body fat, blood pressure, diet questionnaire, physical activity and sociocultural characteristics. For patients with prediabetes and T2DM, the time elapsed since the diagnosis will be obtained, as well as information about pharmacological or non-pharmacological treatment that they are receiving.

For the serological evaluation, a sample of venous blood should be taken in the fasted state, with the aim of measuring the following markers: Fibroblast Growth Factor 21 (FGF21) , Myonectin, and Myostatin. In addition to routine tests such as fasting glycemia, glycosylated hemoglobin, fasting insulinemia, lipid profile (total cholesterol, HDL cholesterol, triglycerides, LDL-C) and C-reactive protein. Additionally, all subjects will participate in an oral glucose tolerance test (OGTT).

In addition to the gold standard of measurement of insulin resistance (hyperinsulinemic-euglycemic clamp), six of the tools currently available for the search of insulin resistance, all derived from calculations from the measurements of The HOMA beta-cell function (HOMA beta-cell%), insulin sensitivity index (ISI), index 1 / fasting insulin, corrected insulin response, insulin / glucose ratio and insulinemia Of fasting.

For each biomarker, an operator / receiver characteristics curve (ROC curve) will be calculated, calculating diagnostic performance and cutoff points with the best combination of sensitivity and specificity. A first approximation will be made to baseline values for these tests, based on the distribution of the tests in healthy, and one or more insulin resistance biomarkers with their recommended cutoff points will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-65 years
* Diligence of informed consent
* Absence of acute illness
* Body mass index less or greater than 25 kg/m2, and presence or absence of a previous diagnosis of diabetes according to the criteria previously stated.

Exclusion Criteria:

* Current therapy with insulin
* Type 1 diabetes
* Oral or injectable anticoagulation
* Previous diagnosis of insulinoma, insulinomatosis, glucagonoma, or other neoplastic disorders of the endocrine pancreas.
* Pregnant women
* BMI <18.5 kg / m2

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults of both sexes, aged between 35 and 65 years, without any significant comorbidity
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2014-08-26 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Incremental area under the insulin curve (iAUCins) | Once in every participant (Cross-sectional). Participants assessed over 6-months
  Area under the insulin curve in a 5-point oral glucose tolerance test, calculated with the trapezoid method, a reliable indicator of whole-body insulin resistance. Expressed in mg*(dL^-1)*(h^-1)
Whole-body glucose disposal | Once in every participant (Cross-sectional). Participants assessed over 6-months
  Glucose disposal when steady state is reached in a hyperinsulinemic-euglycemic clamp, the gold-standard measure of whole-body insulin sensitivity. Expressed in mg*(Kg^-1)*(min^-1)

SECONDARY OUTCOMES:
HOMA-IR (Homeostasis Model Assessment - Insulin Resistance) | Once in every participant (Cross-sectional). Participants assessed over 6-months
  Product of the fasting glycemia in mmol/L and fasting insulinemia in microunits/mL, a surrogate measure of insulin resistance, especially in the fasting state.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos O Mendivil, MD PhD, Principal Investigator — University of Los Andes

IPD SHARING:
Plan to Share IPD: Undecided
Undecided